CLINICAL TRIAL: NCT03762941
Title: Is There a Difference in the Definition and Rating of Quality of Life Among Acute Admitted Elderly i) With and ii) Without Homecare Background: A Cross Sectional Study
Brief Title: Quality of Life Among Acute Admitted Elderly
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-06-2018
Record Dates: First submitted 2018-06-27; First posted 2018-12-04 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Quality of Life
Keywords: Elderly patients; Emergency Department; Homecare
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients acutely admitted: Elderly patients (aged ≥ 65 year) admitted to emergency departments at the Hospital of Southern Jutland or Odense University

SUMMARY:
Elderly dependent on homecare, admitted acutely, are fragile. The aim of this study is to investigate the difference in the definition and rating of Quality of Life (QoL) among acute admitted elderly i) with and ii) without homecare background.

DETAILED DESCRIPTION:
The study is designed as a cross sectional study and will be conducted at three Emergency Departments (ED) within the Region of Southern Denmark; Hospital of Southern Jutland, Hospital of Southwest Jutland and Hospital Lillebaelt. The study method is based on a QoL questionnaire preformed as a structured interview with elderly who are acutely admitted in an ED.

Elderly persons who meet the inclusion criteria will be invited to participate during their admission. Written information about this study will be handed from the nurse in the ED. If the elderly accept she/he will get further oral information from the researcher. Written consent will be obtained if the elderly wish to participate.

Including patients from three different EDs will presumably provide a broad selection, with elderly persons who live both in the city and in rural areas and thereby representing a general sample of the Danish population.There may be a variation in cause of hospitalization related to seasonal changes. To present a broad selection, the inclusion period will involve summer, fall, and winter. Inclusion and all structured interviews will be performed during admission by two persons: the responsible researcher and a research assistant.

Primary Outcome:

The primary outcome QoL will be accessed and evaluated by the Schedule for the Evaluation of Individual Quality of Life - direct weighting (SEIQoL-DW).

Exposure:

Homecare: Receiving "personal" homecare for more than 2 hours per week. Furthermore numbers of hours of homecare a week will be registered for each participant to see if there is any difference in QoL connected to number of hours.

Readmission: Readmissions 30 days after discharge from the primary index admission (yes/no). Readmission is defined as; an unscheduled hospitalization for any reason and where the patient has stayed at the hospital overnight within 30 days after discharge from the index admission.

The outcomes and variables will be collected through;

At a structured interview during hospitalization; The Ph.D student and the research assistant are responsible for conducting the interviews. The patients will at the interview be asked about; Aspect and index score of QoL, cognitive functioning (OMC score), marital status, length of education and social support.

In the patients' records during hospitalization; The Ph.D student is responsibility for collecting following information in the patients' record; Last admission, hours of homecare, use of home nursing, primary reason for hospitalization and comorbidities. Patients will be asked specific for permission to access journal data. Variables from the patients' record will be extracted after the informed consent for participation is obtained. The information from the journal will be handled from health professionals in the ED.

In the patients' record 30 days after discharge; Variables after 30 days will be counted from the discharge form the index admission. The Ph.D student is responsibility for collecting the information in the patient record about readmission and length of hospital stay under the same terms as described above.

Instrument

The primary outcome QoL are accessed and evaluated by SEIQoL-DW which are assessed in a structured interview. First the interviewer elicits five areas of life considered most important by the participant. Secondly, the participant rates the level each of these areas from worst possible to best possible on a visual analogue scale (SEIQoL - VAS) and thirdly the participant is asked for the relative importance of each area by a direct weighting (DW) procedure. The DW procedure uses a pie chart consisting of five coloured segments. Each colour represents an area chosen by the respondent. The areas can be adjusted in size to reflect the relative importance of each area (greatest importance is the largest pie area). The total value of all five segments equals 100. To calculate the participants QoL at the moment, each area will be divided by 100. By multiplying the level of the area by the weight for each area and adding up the values for each area, a SEIQoL-DW index score will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients (aged ≥ 65 year) admitted to EDs at the Hospital of Southern Jutland, Hospital of Southwest Jutland or Hospital Lillebaelt

Exclusion Criteria:

* Patients unable to give informed consent to participate
* Patients known or believed to be cognitively impaired as assessed by the OMC test (score > 18 point).
* Patients who only receive outpatient treatment in the ED will be excluded
* Patients with an inadequate understanding of written and spoken Danish (assessed by the health professionals at the ED).

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly persons who meet the inclusion criteria will be invited to participate during their admission.
Sampling Method: Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Individual Quality of life accessed and evaluated by a structured interview | d) QoL are measured during admission(expected inclusions period: 1 year). Data are reported ½ year after the end of inclusion.
  The primary outcome is QoL measured as an index score (range from 0 [lowest QoL] to 100 [highest QoL]).

CONTACTS AND LOCATIONS:
Overall Officials: Mette Elkjær, Principal Investigator — University of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, The Region of Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elkjaer M, Primdahl J, Mogensen CB, Brabrand M, Gram B. The quality of life of older adults acutely admitted to the emergency department: A cross-sectional study. Nurs Open. 2022 Jul;9(4):2130-2138. doi: 10.1002/nop2.1223. Epub 2022 Apr 30. PMID 35488717